CLINICAL TRIAL: NCT06673212
Title: Barley to Support Food and Drink Innovation (RI-B7-3)
Brief Title: Black Barley Study - Barley to Support Food and Drink Innovation (RI-B7-3)
Acronym: BB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ROW_2022_001
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Wheat Bread (Active Comparator): Control Wheat Bread will be prepared to the same formulation as white wheat bread.
  Interventions: Other: Control Wheat Bread
- Berneray Bere barley bread (Experimental): Berneray Bere barley bread will be prepared to a formulation as for the white wheat bread, but the wheat flour will be replaced with Berneray Bere barley flour.
  Interventions: Other: Berneray Bere barley bread
- Black Barley bread (Experimental): Black Barley bread will be prepared to a formulation as for the white wheat bread, but the wheat flour will be replaced with Black Barley flour.
  Interventions: Other: Black Barley bread

INTERVENTIONS:
Other: Control Wheat Bread — Ingredients: Wheat Flour, Salt, Water, Allinson's Dried Active Yeast, Sugar
  Arms: Control Wheat Bread
Other: Berneray Bere barley bread — Ingredients: Berneray Bere Barley Flour, Salt, Water, Allinson's Dried Active Yeast, Sugar
  Arms: Berneray Bere barley bread
Other: Black Barley bread — Ingredients: Black Barley Flour, Salt, Water, Allinson's Dried Active Yeast, Sugar
  Arms: Black Barley bread

SUMMARY:
Sustained postprandial hyperglycaemia is an independent risk factor for cardiovascular complications and death. Intensive glucose control is the predominant factor to prevent the development of chronic complications in Type 2 Diabetes Mellitus (T2DM). The investigators have shown that phytochemical-rich extracts (in this case anthocyanins and their derivatives) can attenuate glucose response and there is also strong evidence for the role of fibre. Here a selected barley line (rich in anthocyanins and (1,3;1,4)-β-glucan) will be compared to a control barley and control wheat in an acute human dietary intervention (with n=15 healthy volunteers) to explore the potential to modulate postprandial glycaemia and insulinaenemia. An additional secondary outcome will include metabolomics analysis of the blood plasma and urine to detect differences in bioactive compounds including phytochemical metabolites. This will help ensure that barley lines being bred for human food can also deliver benefits for health.

DETAILED DESCRIPTION:
Barley is an important Scottish crop in terms of contributing to the distilling industry but underutilised as a healthy (and potentially sustainable food). The investigators have shown (unpublished data) that barleys entering the food supply chain are not bred for food but are often grain destined for distilling and not rich is components of value for human nutrition, for example (1,3;1,4)-β-glucan, micronutrient vitamins and minerals as well as bioactive phytochemicals associated with reduction of non-communicable diseases such as type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD).

Current research is exploring the potential of specifically bred food barleys to require less inputs in terms of nutrients and pesticides and grow on more marginal lands providing farmers with a crop harvested at a different time of year, mitigating against unpredictable weather and a changing climate. It is important that these barleys also deliver benefits to human health. There are established health claims with regard to the lipid lowering effect of (1,3;1,4)-β-glucan and phytochemical-rich barleys could also potentially reduce blood glucose, an important factor leading to metabolic deregulation and subsequent disease development. This would meet the needs of people choosing a healthy lifestyle, as well as those living with or at risk of T2DM. From the food collections being developed at the James Hutton Institute, an accession (high in (1,3;1,4)-β-glucan and phytochemicals) will be selected and tested in an acute dietary intervention to determine if postprandial blood glucose levels are reduced. This will be compared to control barley and wheat products.

ELIGIBILITY:
Inclusion Criteria:

Apparently healthy male and female subjects with Diabetes Risk Score ≥ 7 points

Exclusion Criteria:

* Type 1 diabetes
* Type 2 diabetes controlled with medication
* Coeliac Disease
* Eating disorders (anorexia, bulimia, binge eating or night eating syndrome)
* Food allergies/intolerances
* Any significant health issues
* Breastfeeding/ Pregnancy
* Addiction to any substances
* Are unable to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose levels | 5 hours
  Modulation of postprandial blood glucose levels after acute consumption of the Black barley, Bere barley and the Wheat breads.
Postprandial insulin levels | 5 hours
  Modulation of postprandial insulin levels after acute consumption of the Black barley, Bere barley and the Wheat breads.

SECONDARY OUTCOMES:
Concentration of phytochemical metabolites in the systemic circulation | 5 hours
  Changes in phytochemical metabolites after acute consumption of the Black barley, Bere barley and the Wheat breads.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Russell, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No